CLINICAL TRIAL: NCT02005861
Title: "One-step" Bone Marrow Mononuclear Cell Transplantation in Talar Osteochondral Lesions
Acronym: BMDC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0008310; 11.03.2013 (Other: Regione Emilia Romagna)
Record Dates: First submitted 2013-11-05; First posted 2013-12-09 (Estimated); Last update posted 2023-05-12 (Actual); Status verified 2017-08

CONDITIONS: Osteochondritis
Keywords: osteochondral lesion; talus; ankle; cartilage repair
MeSH Terms: conditions — Osteochondritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bone marrow cells transplantation (Experimental): surgical procedure :the day before the surgery: platelet gel production. The day of the surgery: bone marrow aspiration from the posterior iliac crest of the patient and concentration. After the bone marrow harvesting, ankle arthroscopy will be performed. The lesion will be detected and cleaned.
  An equine collagen type 1 scaffold (IOR-G1, Novagenit, Mezzolombardo, TN, Italy) will be loaded with 2 ml of bone marrow concentrate and implanted.
  After that platelet gel will be loaded on the top of implant
  Interventions: Procedure: bone marrow cells transplantation on collagen scaffold

INTERVENTIONS:
Procedure: bone marrow cells transplantation on collagen scaffold — 120 ml of venous blood will be collected for the platelet gel production. The day of the surgery, 60 ml of bone marrow will be aspirate from the posterior iliac crest and concentrated. a standard ankle arthroscopy will be performed, with the patient in the supine position. The lesion will be detected and cleaned.
  An equine collagen type 1 scaffold (IOR-G1, Novagenit, Mezzolombardo, TN, Italy) will be loaded with 2 ml of bone marrow concentrate and cut into an appropriate shape to fit the lesion.
  After the scaffold implantation 2 ml of platelet gel will be loaded on the top of implant, in order to provide growth factors and to improve the stability of the implant.
  Other Names: kit IOR-G1, a collagen scaffold; Autologous platelet gel will be implanted on the scaffold

SUMMARY:
BACKGROUND Osteochondral lesions are defects of the cartilaginous surface and underlying subchondral bone of the talar dome.

The use of concentrated bone marrow derived cells has been gaining successful results with arthroscopic implantation, since it is possible to transplant not only mesenchymal stem cells but also accessory cells that support angiogenesis and vasculogenesis by producing several growth factors.

OBJECTIVES Objective of this project is to identify the critical points of the regenerative treatment of osteochondral lesions of the ankle, in order to develop a standard and predictable procedure able to overcome the drawbacks of the previous techniques.

METHODS Our program is to evaluate and follow 140 new patients with focal osteochondral lesion of the talus. The surgical procedure will be executed as following: the day before the surgery the platelet gel will be produced. The day of the surgery bone marrow will be aspirate from the posterior iliac crest and concentrated directly in the operating room by centrifugation, in order to obtain 6 mL of concentrate containing nucleated cells.

Then a standard ankle arthroscopy will be performed. The scaffold will be loaded with 2 ml of bone marrow concentrate and cut into an appropriate shape.

After the scaffold implantation platelet gel will be sprayed on the top of implant, in order to provide extra growth factors and to improve the stability of the implant.

All patients will be examined clinically preoperatively, at 3, 6, 12, 24 and 36 months and at maximum follow-up. Different score scales will be used to objectivate the clinical results (AOFAS, SF-36, VAS). X-rays and MRI scan will be also taken preoperatively, and MRI will be executed at 12, 24 and 36 months of follow-up. In particular, a new qualitative MRI called T2 mapping will be performed at 24 months.

EXPECTED RESULTS We expect to highlight the effectiveness of the arthroscopic bone marrow derived cells (BMDCs) transplantation in a long term follow up study, with particular attention to identify the patient population that can gain the maximum benefit from this treatment, avoiding expensive and unnecessary procedures that too often are performed.

DETAILED DESCRIPTION:
Study design The study will be an observational prospective study. 46 patients previously operated in our center by Autologous Chondrocyte Implantation (ACI) will be used as control.

Patients 140 patients with osteochondral lesions of the talar dome will be recruited for this study. All the procedures will be performed according with specific European and Italian guidelines.

The patients will be operated as inpatients in the II Clinic of Orthopaedics and Traumatology. This is an highly specialized ward for the treatment of foot and ankle diseases. During the first day of hospitalization the patients will undergo a complete blood test and standard X-rays examination, along with specialized anesthesiologist, hematological and orthopaedic examinations.

Key inclusion and exclusion criteria Patients must satisfy the following inclusion criteria: osteochondral lesions of the talar dome ICRS grade III or IV lesion, size of the lesion >1.5 cm2, age <50 years.

Key exclusion criteria will take into account the presence of arthritis, kissing lesions, ankle malalignment and ankle instability, articular infections, hematological or rheumatic disorders.

Treatment The surgical procedure will be executed as following: the day before the surgery 120 ml of venous blood will be collected for the platelet gel production performed with an automatic method by Unit 5. The day of the surgery, 60 ml of bone marrow will be aspirate from the posterior iliac crest of the patient and concentrated directly in the operating room by a specific device (kit IOR-G1, Novagenit, Mezzolombardo, TN, Italy), in order to obtain 6 mL of concentrate bone marrow (CBM) containing nucleated cells (stem cells, monocytes, lymphocytes, and other bone marrow resident cells). After the bone marrow harvesting phase, a standard ankle arthroscopy will be performed, with the patient in the supine position. The lesion will be detected and cleaned.

An equine collagen type 1 scaffold (IOR-G1, Novagenit, Mezzolombardo, TN, Italy) will be loaded with 2 ml of bone marrow concentrate and cut into an appropriate shape to fit the lesion.

After the scaffold implantation 2 ml of platelet gel will be loaded on the top of implant, in order to provide growth factors and to improve the stability of the implant.

Patient will be hospitalized for 2 days after surgery. Examinations, MRI and X-rays will be performed in ambulatory in outpatients regimen at the outpatients facility of Rizzoli Orthopaedic Institute.

The evaluation of the different growth factors present in bone marrow releasate was also performed in order to highlight the differences among patient samples.

Statistical analysis (Potency) with calculation Continuous data will be described as means and standard deviations. Qualitative data will be expressed as frequencies and percentages. The Kolmogorov-Smirnov test will be used to evaluate the normality of data distribution. The Levene test will be used to analyze the homoscedasticity. Differences between preoperative and follow up data will be evaluated with the paired t test for homoscedastic and normally distributed data; otherwise, the nonparametric Wilcoxon-Mann-Whitney test will be used. Differences between groups will be evaluated with the unpaired t test for homoscedastic and normally distributed data; otherwise, the nonparametric Wilcoxon-Mann-Whitney test will be used. Pearson's correlation will be performed to investigate the relationships between continuous variables if they will be both normally distributed; otherwise, the Spearman rank correlation test will be used. Statistical analysis will be performed using SPSS® software (Version 15.0; SPSS Inc, Chicago, IL).

Ethical aspect All the patients, in order to be enrolled in this study, must sign a specific informed consent, approved from an independent ethical committee.

Risk for patients Risk for the patients will be the risk related to the surgical procedure. They include anesthetics (local or general), procedure-related risk such as infection, deep venous thrombosis, damages of anatomical structures. It is important to underline that all these risks are not specifically related with this procedure, but with all the procedures involving an ankle arthroscopy with cartilage treatment. The risks for the patients will be minimized with specific training activities for all the personnel taking part to the project (i.e nurses, operating room personnel, attending surgeons, hematologists, residents) . Data will be evaluated by a statistician , and all the monitoring activities will be performed by dedicated personnel.

Good clinical practice For each patient entered into the study a Case Record Form (CRF) in compliance with Good Clinical Practice will prepared. This document does not coincide with the subject's clinical personal folder. It must be given all the data elements relevant to the study. The coordinator of the trial will provide a CFR copy in electronic format to the PU involved. The compilation and maintenance of CRF as well as data transmission to the scientific director of the WP are under the responsibility of the leader of the PU involved.

Patient data will be collected in dedicated databases (on special software) that will enable safe storage and processing, to ensure the privacy of patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Osteochondral lesions of the talar dome
* Presence of lesion classified as ICRS grade III or IV
* size of the lesion >1.5 cm2
* age <50 years

Exclusion Criteria:

* Presence of osteoarthritis
* presence of concomitant tibial lesion
* presence of ankle malalignment
* presence of ankle instability
* presence of rheumatic diseases

Ages: 13 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Estimated)
Dates: Start 2013-04 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
American Orthopaedic Foot and Ankle Society hindfoot score | 24 months after surgery
  American Orthopaedic Foot and Ankle Society hindfoot score will be used to assess the quality of life of the patients with a minimum score of 0 and a maximum of 100.

SECONDARY OUTCOMES:
T2 mapping MRI value | 12 and 24 months after surgery
  MRI will be performed with T2 mapping sequences and T2 values will be recorded as indicator of quality through water content of the regenerated tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Giannini, Prof, Principal Investigator — Rizzoli Orthopaedic Institute, Bologna, Italy
Locations (1):
- I Clinic, Rizzoli Orthopaedic Institute, Bologna, Italy